CLINICAL TRIAL: NCT00965133
Title: Enthusiasm - Sweat - Satisfaction! In Youngster With CP
Brief Title: Endurance Training in Young Persons With Cerebral Palsy; Evaluation of Training Method and Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reidun Lauglo (Other)
Collaborators: Rosenborgklinikken (Unknown); Norwegian University of Science and Technology (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Reidun Lauglo, Physiotherapist, Reidun Lauglo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shdir-08/4914
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Normal daily activity (No Intervention)
  Interventions: Other: Endurance training intervention

INTERVENTIONS:
Other: Endurance training intervention — High intensive interval training of walking / running on treadmill for 1 1/2 - 4 minute,repeated minimum 4 times, at an intensity equalling at least 80% of maximal heart frequency. Performed 2-5 times per week for 4-8 weeks, totally 24 sessions.

SUMMARY:
The hypotheses of the study are that children / youth with CP will by possibly use of technical aids be able to perform high intensity endurance training by walking / running on a treadmill, and that this training will improve their health by increased aerobic capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Person with CP, GMFCS-level I-IV, age 10-17 years
* Living in Mid-Norway
* Wants to increase his / her level of physical activity

Exclusion Criteria:

* Completes less than 75% of the total number of training sessions
* Not able to complete the testing and training procedures due to sickness, injury or other physical and psychological conditions

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity | Sept. 2009 - april 2010

SECONDARY OUTCOMES:
Quality of life | Sept. 2009 - April 2010

CONTACTS AND LOCATIONS:
Locations (1):
- Rosenborgklinikken, Trondheim, Norway

REFERENCES:
- [Derived] Lauglo R, Vik T, Lamvik T, Stensvold D, Finbraten AK, Moholdt T. High-intensity interval training to improve fitness in children with cerebral palsy. BMJ Open Sport Exerc Med. 2016 May 9;2(1):e000111. doi: 10.1136/bmjsem-2016-000111. eCollection 2016. PMID 27900177